CLINICAL TRIAL: NCT05492214
Title: The Effect of Time Window for Umbilical Cord Clamping During Cesarean Section on the Health Outcomes of Offspring Hemoglobin and Maternal Blood Loss
Brief Title: The Effect of Time Window for Umbilical Cord Clamping During Cesareans on Offspring Hemoglobin and Maternal Blood Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Liuyang Maternal and Child Health Care Hospital (Unknown); Women and Children's Health Care Hospital of Huantai (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NSFC.82173528
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Delayed Cord Clamping; Hemoglobin; Blood Loss
Keywords: Cesarean delivery; Time window for umbilical cord clamping; Maternal and neonatal health outcome; Anemia; Randomized controlled trial
MeSH Terms: conditions — Hemorrhage; Anemia | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Delay 30s group (Experimental): Cord clamping will be delayed at 30 seconds after delivery.
  Interventions: Procedure: Delayed cord clamping (30s)
- Delay 60s group (Experimental): Cord clamping will be delayed at 60 seconds after delivery.
  Interventions: Procedure: Delayed cord clamping (60s)
- Delay 90s group (Experimental): Cord clamping will be delayed at 90 seconds after delivery.
  Interventions: Procedure: Delayed cord clamping (90s)
- Control group (No Intervention): Cord clamping will be immediate (within 15 seconds) after delivery, in accordance with the standard practice in the study sites

INTERVENTIONS:
Procedure: Delayed cord clamping (30s) — The same as that stated in arm descriptions.
  Arms: Delay 30s group
Procedure: Delayed cord clamping (60s) — The same as that stated in arm descriptions.
  Arms: Delay 60s group
Procedure: Delayed cord clamping (90s) — The same as that stated in arm descriptions.
  Arms: Delay 90s group

SUMMARY:
This is a randomized controlled trial, aiming to evaluate the effects of time window for umbilical cord clamping during cesarean section on the health outcomes of offspring hemoglobin，maternal blood loss，and children's growth and development. It will be conducted in Liuyang city and Huantai county of China, and the targeted sample size is 360 (180 in each site). All the eligible pregnant women will be randomly assigned to one of the four groups (three intervention groups and one control group), and their babies will be followed up to 18 months of age.

DETAILED DESCRIPTION:
The World Health Organization and American College of Obstetricians and Gynecologists have recommended a delay in umbilical cord clamping after birth, irrespective of delivery modes, which was based on studies from vaginal deliveries rather than cesareans. In cesareans, the optimal time window for umbilical cord clamping has not been determined, and the relevant safety data are limited. In this randomized study, the investigators aim to evaluate the impacts of time window for umbilical cord clamping during cesarean section on maternal and child health outcomes, and to evaluate the optimal timing of the clamping. The investigators are planning to enroll 360 pregnant women scheduled for cesareans, and to randomly allocate them into four groups: the umbilical cord will be clamped within 15 seconds (immediately), or delayed after deliveries for 30, 60, and 90 seconds, respectively. Babies will be followed up at 3, 6, 12, and 18 months of age. Maternal hemoglobin before and after cesareans, neonatal hemoglobin, children's hemoglobin at 6, 12, 18 months of age will be measured. At each follow-up visit, children's length and weight will be measured, their development will be assessed, and a questionnaire survey including information on feeding, sleep, and medication will be conducted. The primary outcomes are the neonatal hemoglobin and the change in maternal hemoglobin. The secondary outcomes include the incidence rate of neonatal anemia and jaundice, Apgar score, the incidence rate of neonatal intensive care unit (NICU) admission, placental weight, maternal hemoglobin after the cesarean, estimated maternal blood loss, and the incidence rate of maternal blood transfusion. In addition, the children's hemoglobin, anemia, growth and development are considered as the exploratory secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* local resident in Liuyang city, Huantai county and their surrounding areas
* Singleton pregnancy
* Elective caesarean, or cesarean section after the start of labor but the cervix is less than 3 cm
* Term pregnancy (≥37 weeks of gestation), and the fetal weight was estimated ≥2500g by intrauterine ultrasound
* Written informed consent is obtained

Exclusion Criteria:

* Pregnant women with the following risk factors: severe hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥110mmHg), preeclampsia, chronic hypertension with preeclampsia, diabetes mellitus with severe microangiopathy, placenta previa, placenta implantation, placental abruption, intrauterine distress, prenatal infection, severe anemia (hemoglobin<7g/dL), coagulation disorders, thrombosis disease
* Plan to retain cord blood
* Rh-negative pregnant women
* Prenatal diagnosis of fetal abnormalities which may lead to difficulties in cesareans or adverse pregnancy outcomes, such as abnormal heart monitoring, fetal distress, malformation, anemia, and intrauterine growth restrictions
* Other conditions not suitable for intervention as judged by obstetricians

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The neonatal hemoglobin | Within 72 hours after birth
  In the heel blood
The change in maternal hemoglobin | Within 72 hours before the cesarean, and within 72 hours after the cesarean
  Difference in maternal hemoglobin levels before and after the cesarean

SECONDARY OUTCOMES:
The incidence rate of neonatal anemia | Within 72 hours after birth
  Defined as hemoglobin <145g/L
The incidence rate of neonatal jaundice | Before discharging from hospitals, usually within 1 week after birth
  The incidence rate of neonatal jaundice
Apgar score | At 1 min, 5 min, and 10 min after birth
  An indicator for the activity, pulse, grimace, appearance, and respiration of neonates. It ranges from 0 to 10, the higher the better.
The incidence rate of neonatal intensive care unit admission | Before discharging from hospitals, usually within 1 week after birth
  The incidence rate of neonatal intensive care unit admission
Placental weight | At birth
  In grams
Maternal hemoglobin after the cesarean | Within 72 hours after the cesarean
  In venous blood
Estimated maternal blood loss | During the cesarean
  By volume-method and area-method
The incidence rate of maternal blood transfusion | At delivery
  The incidence rate of maternal blood transfusion

OTHER OUTCOMES:
The children's hemoglobin | At 6, 12, 18 months of age
  In fingertip blood
The children's anemia | At 6, 12, 18 months of age
  Defined as hemoglobin <110 g/L
The children's length | At 3, 6, 12, 18 months of age
  In Z-score
The children's weight | At 3, 6, 12, 18 months of age
  In Z-score
The results of Denver Developmental Screening Test | At 3, 6, 12, 18 months of age
  The abnormal rate

CONTACTS AND LOCATIONS:
Overall Officials: Jianmeng Liu, Principal Investigator — Peking University; Hongtian Li, Study Director — Peking University
Locations (2):
- China (2):
  - Liuyang Maternal and Child Health Care Hospital, Guankou, Hunan
  - Women and Children's Health Care Hospital of Huantai, Zibo, Shandong

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared upon the request of other researchers, and all the key variables that will be reported in the main paper are planned to be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After the publication of the main paper (hopefully before the end of 2024), the data will be available to share to other researchers
Access Criteria: Researchers should request the data via the following Email: lihongtian@pku.edu.cn or liujm@pku.edu.cn

REFERENCES:
- [Derived] Song Q, Li H, Mu Y, Xiong Y, Liu Y, Liu Y, Jin C, Huang X, Zhao L, Zhang M, Zhou Y, Liu J. Effects of Delayed Umbilical Cord Clamping at Different Timings on Neonatal Hemoglobin and Maternal Blood Loss During Cesarean Delivery at Term: A Randomized Controlled Trial. J Pediatr. 2025 Aug;283:114620. doi: 10.1016/j.jpeds.2025.114620. Epub 2025 Apr 23. PMID 40280473

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT05492214/SAP_000.pdf